CLINICAL TRIAL: NCT00697697
Title: A Randomized, Double-blind, Active-controlled, Phase 3 Extension Study Investigating the Safety and Efficacy Over 40 Weeks of 2 Doses of MAP0010 in Asthmatic Children (12 Months to 8 Years Old at the Time of Enrollment Into the MAP0010-CL-P301 Study)
Brief Title: A Study of 2 Doses of MAP0010 in Asthmatic Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporate decision
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAP0010-CL-P301X
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2013-10-23 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: asthmatic children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.135mg MAP0010 (Experimental): 0.135mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 40 weeks
  Interventions: Drug: 0.135mg MAP0010
- 0.25mg MAP0010 (Experimental): 0.25mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 40 weeks
  Interventions: Drug: 0.25mg MAP0010

INTERVENTIONS:
Drug: 0.135mg MAP0010 — 0.135mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 40 weeks
  Arms: 0.135mg MAP0010
Drug: 0.25mg MAP0010 — 0.25mg MAP0010 (unit dose budesonide) delivered by nebulization twice daily for 40 weeks
  Arms: 0.25mg MAP0010

SUMMARY:
The purpose of this study is to examine the safety of two doses of MAP0010 in asthmatic children, 12 months to 8 years of age, over a 40-week period.

ELIGIBILITY:
Inclusion Criteria:

* Completed 12 weeks of treatment in the MAP0010-CL-P301 study.
* Patient, parent, and guardian (as appropriate) are willing for child to undergo all study procedures and willing to sign the informed consent and assent, as appropriate.

Exclusion Criteria:

* Less than 80% compliance with either study treatment and/or other study procedures (e.g., completion of symptom e-diary) in the MAP0010-CL-P301 Study.

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MAP Pharmaceuticals

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.135mg MAP0010 | 0.25mg MAP0010
Started | 94 | 98
Completed | 45 | 44
Not Completed | 49 | 54

BASELINE CHARACTERISTICS:
Population: Subjects were randomly assigned to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.135mg MAP0010 | 0.25mg MAP0010 | Total
Number analyzed (Participants) | 94 | 98 | 192
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.6 (2.50) | 4.9 (2.03) | 4.8 (2.27)
Age, Continuous [Median (Full Range); unit: years] | 5.0 [1 to 9] | 5.0 [1 to 8] | 5.0 [1 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 37 | 83
  Male | 48 | 61 | 109

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events Related to Study Drug
Description: A treatment emergent adverse event is one with a start date on or after the date of first administration of the study drug during the study.
Time Frame: 40 weeks
Population: All patients who received any study drug and who had at least one post safety evaluation were included in the adverse event analysis.
Measure: Number; unit: participants
Arm/Group | 0.135mg MAP0010 | 0.25mg MAP0010
Number analyzed (Participants) | 94 | 98
participants | 6 | 4

2. Primary Outcome: Number of Patients Reporting at Least One Treatment Emergent Adverse Event Leading to Study Termination
Description: as for outcome 1
Time Frame: 40 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 0.135mg MAP0010 | 0.25mg MAP0010
Number analyzed (Participants) | 94 | 98
participants | 8 | 7

ADVERSE EVENTS:
Description: All patients who received any study drug and who had at least one post safety evaluation were included in the adverse event analysis.
Arm/Group | 0.135mg MAP0010 | 0.25mg MAP0010
Serious Adverse Events (participants affected / at risk) | 0/94 | 1/98
Other Adverse Events (participants affected / at risk) | 71/94 | 85/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.135mg MAP0010 (N=94) | 0.25mg MAP0010 (N=98)
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.135mg MAP0010 (N=94) | 0.25mg MAP0010 (N=98)
Pyrexia (General disorders) | 4 | 12
Pharyngitis (Infections and infestations) | 2 | 6
Pharyngitis streptococcal (Infections and infestations) | 10 | 5
Rhinitis (Infections and infestations) | 2 | 5
Sinusitis (Infections and infestations) | 7 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 17 | 32
Viral Infection (Infections and infestations) | 3 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Gastritis (Gastrointestinal disorders) | 1 | 5
Nasopharyngitis (Infections and infestations) | 5 | 4
Otitis Media (Infections and infestations) | 4 | 5

LIMITATIONS AND CAVEATS:
The study was terminated due to a corporate decision before all subjects had completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.